CLINICAL TRIAL: NCT00644683
Title: A Pilot Observational Study to Assess Changes in Biochemical Parameters of Ovarian Reserve With Chemotherapy
Status: Completed | Type: Observational
Sponsor: Lynn Henry (Other)
Responsible Party: Sponsor-Investigator, Lynn Henry, Principal Investigator, University of Michigan Rogel Cancer Center
Organization: University of Michigan Rogel Cancer Center (Other)
Other Study IDs: UMCC 2007.081; HUM 00014246 (Other: University of Michigan)
Record Dates: First submitted 2008-01-17; First posted 2008-03-27 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: premenopausal women with breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Premenopausal women who are diagnosed with breast cancer are frequently treated with chemotherapy. Chemotherapy can affect the ovaries, and the effects can range from temporary loss of menstrual periods to permanent menopause. It is difficult to predict how an individual's ovarian function will be affected by chemotherapy. There are a number of hormones which can be measured in the blood which are related to fertility and ovarian function. The levels of these hormones may change with chemotherapy, and may relate to the effect of chemotherapy on the ovaries.

In this study, we plan to enroll 28 women ranging in age from 25 to 50 who are diagnosed with breast cancer and will be treated with chemotherapy. We will check blood levels of the hormones before, immediately after, and 1 year after treatment with chemotherapy. We will only be checking these blood tests for this study; the type of chemotherapy given will be up to the patient and her oncologist. We will also ask some questions about factors that can influence the levels of these hormones, such as number of children, age of menopause of other family members, and smoking history. The results from this study will be used to help us develop future studies looking at changes in ovarian function with chemotherapy, and the effects of other breast cancer therapies, such as endocrine therapy, on the ovaries.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be women with a histologically confirmed invasive adenocarcinoma of the breast (stage I, II, or III) with no evidence of metastatic disease.
* Patients must be planning to receive neoadjuvant or adjuvant chemotherapy. Patients may receive concurrent trastuzumab as indicated. If a patient has not yet undergone final surgical resection, it must be highly likely (but is not required to be definite) that the patient will be treated with adjuvant chemotherapy.
* Patients must have:

  * Reached their 25th birthday and not yet reached their 51st birthday at the time of study enrollment, AND
  * Had menses within 3 months prior to starting chemotherapy
* Patients must not have received prior cytotoxic chemotherapy for any oncologic, rheumatologic, or dermatologic condition.
* Patients must not have had prior bilateral oophorectomy or pelvic radiation, and must not have had prior hysterectomy
* ECOG performance status 0 - 2
* Pregnant or nursing women may not participate. Women of reproductive potential must agree to use an effective non-hormonal contraceptive method, such as condoms, tubal ligation, non-hormonal intrauterine device, partner sterilization, and abstinence during chemotherapy.
* All patients must be informed of the investigational nature of this study and given written informed consent in accordance with institutional and federal guidelines.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: premenopausal women with invasive adenocarcinoma of the breast between the ages of 25 and 50.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2007-09; Primary Completion 2012-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
estimates of serum concentrations | 1 year
  To generate estimates of serum concentrations of inhibin A, inhibin B, and anti-Mullerian hormone in premenopausal breast cancer patients (25-50 years of age) before, immediately after, and 1 year following completion of chemotherapy.
  Hypothesis: Serum concentrations of hormones involved in the hypothalamic-pituitary-ovarian axis (anti-Müllerian hormone, inhibin A, inhibin B, and follicle stimulating hormone) are detectable in the serum of all premenopausal women prior to chemotherapy

SECONDARY OUTCOMES:
serum concentrations of reproductive hormones | 1 year
  To determine serum concentrations of reproductive hormones (estradiol and its metabolites) before, immediately after, and 1 year following completion of chemotherapy using standard estradiol assays, and compare these results to those obtained using metabolomics.
  Hypothesis: Serum concentrations of reproductive hormones (estradiol and its metabolites) will be detectable in all premenopausal women before chemotherapy, and will decrease immediately after chemotherapy in a considerable subset of patients. In addition, metabolomics will provide the same information about the presence or absence of estrogens, and will also provide additional data about other compounds present in the serum.
  2

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Henry NL, Xia R, Schott AF, McConnell D, Banerjee M, Hayes DF. Prediction of postchemotherapy ovarian function using markers of ovarian reserve. Oncologist. 2014 Jan;19(1):68-74. doi: 10.1634/theoncologist.2013-0145. Epub 2013 Dec 6. PMID 24319018